CLINICAL TRIAL: NCT04136119
Title: A Survey of Practice of Micronutrient Supplementation in Critically Ill Patients
Brief Title: Micronutrients in Critically Ill Patients
Acronym: MiNuCrit
Status: Completed | Type: Observational
Sponsor: Guy's and St Thomas' NHS Foundation Trust (Other)
Responsible Party: Sponsor
Other Study IDs: IRAS 268780
Record Dates: First submitted 2019-10-21; First posted 2019-10-23 (Actual); Last update posted 2021-03-16 (Actual); Status verified 2019-10

CONDITIONS: Nutrition; Critical Illness; Vitamin Supplementation
Keywords: micronutrient supplementation; vitamins
MeSH Terms: conditions — Critical Illness | interventions — Surveys and Questionnaires

STUDY DESIGN:
Observational Model: Other | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- healthcare professionals: doctors, pharmacists and dieticians who are involved in prescribing vitamins and micronutrients to critically ill patients
  Interventions: Other: questionnaire

INTERVENTIONS:
Other: questionnaire — survey exploring practice of vitamin and micronutrient supplementation

SUMMARY:
Nutritional support is an important component of modern critical care. The practice of vitamin and micronutrient supplementation is variable and official guidelines are not consistent. The primary objective of this observational study is to investigate the clinical practice of micronutrient supplementation during critical illness and to explore the factors underpinning clinical decisions.

DETAILED DESCRIPTION:
Nutritional support is an integral component of modern critical care. Malnutrition is common, but measurement of serum concentrations of most vitamins and micronutrients does not form part of routine care for most critically ill adults in the UK. When measured in a research setting, a large proportion of critically ill patients have low serum concentrations of many essential nutrients. Nutrient deficiency is associated with adverse outcomes, including delirium and increased mortality. To date, it is unclear whether there is a role for micronutrient supplementation in critically ill patients. Official guidelines from the European Society of Parenteral and Enteral Nutrition (ESPEN), American Society of Parenteral and Enteral Nutrition (ASPEN), German Intensive Care Society and Kidney Disease Improving Global Outcome (KDIGO) vary and are contradictory to some extent. Additionally, vitamins B1 and C have been administered as an intervention in the treatment of septic shock and other disease states, but methodological flaws with such studies have left many clinicians with equipoise over the place of vitamin and micronutrients in clinical practice.

There is a need for a well designed, adequately powered intervention study. In preparation, we would like to explore current practice and decision making of doctors, pharmacists and dieticians who are directly involved in prescribing nutritional support.

The primary objective of this observational study is to investigate the clinical practice of micronutrient supplementation during critical illness and to explore the factors underpinning clinical decisions.

ELIGIBILITY:
Inclusion Criteria:

* healthcare professional who is involved in prescribing vitamins or micronutrients to critically ill patients in the ICU

Exclusion Criteria:

* none

Sex: All | Healthy Volunteers: Yes
Age Groups: Child, Adult, Older Adult
Study Population: health care professionals working in the ICU
Sampling Method: Non-Probability Sample
Enrollment: 60 (Actual)
Dates: Start 2019-11-18 (Actual); Primary Completion 2020-02-01 (Actual); Study Completion 2020-12-01 (Actual)

PRIMARY OUTCOMES:
clinical practice of vitamin supplementation | October 2019 - April 2020
  indications for vitamin supplementation
clinical practice of micronutrient supplementation | October 2019 - April 2020
  indications for micronutrient supplementation

CONTACTS AND LOCATIONS:
Locations (1):
- Guy's & St Thomas Foundation Hospital, London, United Kingdom

IPD SHARING:
Plan to Share IPD: No
individual participant data will not be made available